CLINICAL TRIAL: NCT05255913
Title: Effectiveness of Nano-silver Fluoride and Silver Diamine Fluoride for Arresting Early Childhood Caries (a Randomized Clinical Trial)
Brief Title: Effectiveness of Nano-silver Fluoride and Silver Diamine Fluoride for Arresting Early Childhood Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maryam Quritum, dentist, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0265-07/2021
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Early Childhood Caries
Keywords: Caries arrest, early childhood caries, Nanosilver fluoride
MeSH Terms: interventions — colloidal silver; silver diamine fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental)
  Interventions: Drug: Nanosilver
- group 2 (Active Comparator)
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Nanosilver — preventive material for arresting caries
  Arms: group 1
Drug: Silver diamine fluoride — preventive material for arresting caries
  Arms: group 2

SUMMARY:
Aim of the study: To evaluate and compare the clinical cariostatic efficacy of NSF with 38% SDF solution after sex and twelve months in arresting ECC lesions.

The Null hypothesis will be that no statistically significant difference will be detected between the two groups in the arrest of carious lesions in children with ECC.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 4 years old.
* The presence of at least one active carious lesion on a primary tooth, with scores 3 and higher (according to the International Detection and Assessment System- ICDAS II)
* Completion of an informed consent to participate in the study.

Exclusion Criteria:

* Children reporting spontaneous or elicited pain from caries or showing any signs of pulpal infection, swelling and/or abscess, obvious discoloration of the tooth and premature hypermobility.

  * Parental refusal to participate in the study.
  * Allergy or sensitivity to silver or any of the materials included in the study.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
caries arrest | 6 months and 1 year
  percentage of arresting caries in primary teeth

SECONDARY OUTCOMES:
Comparing parental satisfaction and adverse effects with interventions | 6 months
  assessed by a self-rated questionnaire with responses on a 4-point Likert scale ranging from very satisfied, satisfied, unsatisfied, to very unsatisfied - Parents were also asked about adverse effects
Evaluating oral health related quality of life of children and their families. | 6 months and 1 year
  by using the Arabic version of the Early Childhood Oral Health Impact Scale (A-ECOHIS)
Assessing caries increment on remaining teeth in the oral cavity other than the tooth/ teeth receiving the preventive agent | 6 months and 1 year
  caries increment which is the number of new caries lesions developed over the study period detected using dmfs (change in dmfs score)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Quritum M, Abdella A, Amer H, El Desouky LM, El Tantawi M. Effectiveness of nanosilver fluoride and silver diamine fluoride in arresting early childhood caries: a randomized controlled clinical trial. BMC Oral Health. 2024 Jun 18;24(1):701. doi: 10.1186/s12903-024-04406-3. PMID 38890627
- [Derived] Quritum M, Abdella A, Amer H, El Tantawi M. Effect of silver diamine fluoride and nano silver fluoride on oral health-related quality of life of children with early childhood caries: A randomized clinical trial. J Dent. 2024 Mar;142:104878. doi: 10.1016/j.jdent.2024.104878. Epub 2024 Feb 2. PMID 38311016